CLINICAL TRIAL: NCT05146076
Title: Home-based Physical Trainings for Reducing Cardiovascular Risk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: István Kósa (Other)
Responsible Party: Sponsor-Investigator, István Kósa, Head of Department of Medical Prevention, Szeged University
Organization: Szeged University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CV risk physical training
Record Dates: First submitted 2021-10-19; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telemedicine supervised group (Experimental): physical training supervised by telemonitoring
  Interventions: Other: home-based physical training
- institutional training (Active Comparator): institutional training supervised by physiotherapist
  Interventions: Other: institutional physical training

INTERVENTIONS:
Other: home-based physical training — home-based physical training minimum 150 min./week with telemonitoring
  Arms: telemedicine supervised group
Other: institutional physical training — institutional physical training supervised by physiotherapist 2-3 times 60 min./week
  Arms: institutional training

SUMMARY:
Prospective intervention study among metabolic syndrome patients, investigating the effects of 12 weeks home-based physical training programme with telemonitoring on the anthropometric parameters, the exercise tolerance and other cardio-metabolic risk factors of the metabolic syndrome.

DETAILED DESCRIPTION:
Prospective intervention study among metabolic syndrome patients, investigating the effects of 12 weeks home-based physical training programme with telemonitoring on the anthropometric and laboratory parameters, the exercise tolerance and other cardio-metabolic and other psycho-social (anxiety, depression, vital exhaustion , sleep disturbances) risk factors of the metabolic syndrome.

ELIGIBILITY:
Inclusion criteria:

* voluntary patients aged between 25 and 70 years
* low level of regular physical activity, less than 30 min./ week
* basic IT skills
* 3 risk factors present out of the 5 metabolic risk factors from the followings:

  1. waist circumference (WC) above 102 cm in men and above 88 cm in women
  2. proved type 2 diabetes mellitus (T2DM) or fasting plasma glucose level above 5,6 mmol/l
  3. treated hypertension or spontaneous blood pressure higher or equivalent than 130/ 85 mmHg
  4. treated hypertriglyceridaemia or serum triglyceride level above 1,7 mmol/l
  5. serum HDL cholesterol level under 1,03 mmol/l in men or 1,3 mmol/l in women

Exclusion Criteria:

* any upcoming planned invasive cardiological intervention
* uncontrolled hypertension
* type one diabetes mellitus (T1DM)
* T2DM which needed more than 1 dose insulin per day
* chronic heart failure
* chronic renal failure
* serious cognitive disfunction
* lack of cooperation
* any of known disease or condition that seriously affect the mental and legal capacity
* any other conditions inhibiting regular physical trainings

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
waist circumference (WC) navel | 12 weeks
  waist circumference measured at navel level
Six minutes walk distance (6MWD) | 12 weeks
  6 minutes walk distance

SECONDARY OUTCOMES:
body parameter 1 | 12 weeks
  body weight measured in kg-s
body parameter 2 | 12 weeks
  hip circumference measured in cm-s
body parameter 3 | 12 weeks
  BMI calculated from weight (kg-s) and height (m-s)
body parameter 4 | 12 weeks
  body composition parameters (fat / muscle / water ratio)
functional parameter 1 | 12 weeks
  stress ECG duration time measured in sec
laboratory parameter 1 | 12 weeks
  glycated haemoglobin (HbA1c) measured in percentage
laboratory parameter 2 | 12 weeks
  fasting plasma glucose (+PG) measured in mmol/l
laboratory parameter 3 | 12 weeks
  triglyceride (TG), measured in mmol/l
laboratory parameter 4 | 12 weeks
  HDL cholesterol, measured in mmol/l
laboratory parameter 5 | 12 weeks
  total-cholesterol measured in mmol/l
psychological test result 1 | 12 weeks
  Anxiety score
psychological test result 2 | 12 weeks
  Depression score
psychological test result 3 | 12 weeks
  vital exhaustion score
psychological test result 4 | 12 weeks
  health locus of control score
psychological test result 5 | 12 weeks
  perceived stress score
psychological test result 6 | 12 weeks
  self-control score

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged, Faculty of Health Sciences and Social Studies, Department of Phisiotherapy, Szeged, Hungary